CLINICAL TRIAL: NCT04185727
Title: Training Intervention in the Treatment of Anorexia Nervosa (STRONG_2)
Brief Title: Training Intervention in the Treatment of Anorexia Nervosa
Acronym: STRONG_2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Corona.
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other); University of South-Eastern Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-19037864
Record Dates: First submitted 2019-11-12; First posted 2019-12-04 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2019-11

CONDITIONS: Anorexia Nervosa; Exercise
Keywords: feeding and eating disorders; training; supervised exercise; muscle strength; anorexia nervosa; bone health; psychopathology; pathophysiology; intervention; prospective
MeSH Terms: conditions — Anorexia Nervosa; Motor Activity; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled open trial, comparing the effect of Standard of care (SOC) with Standard of care + strength training.
  The interventional clinical trial design includes two parallel groups and 12 weeks exposure. The goal is to include 24-30 patients.
  The study will allocate patients to groups consisting of 4 members who receive either SOC or SOC + strength training for 12 weeks. All participants are assessed at baseline, after 1 week, after 6 weeks, post-treatment (12 weeks), and at 6 months' post follow-up (24 weeks) and monitored for changes in physiological, biological and psychological variables. Some tests are also done more frequently. The strength training program will consist of three weekly supervised strength exercise sessions, each 40-60 min of duration, which starts with a 10 min warm-up and are completed with a meditation/relax session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Therapy control group
- Standard of Care (SOC) + strength training (Experimental): Strength training intervention as add on to therapy
  Interventions: Other: Supervised strength training

INTERVENTIONS:
Other: Supervised strength training — 12 weeks supervised strength training exposure. The study will allocate patients to groups consisting of 4 members who receive strength training for 12 weeks. The strength training program will consist of three weekly supervised strength exercise sessions, each 40-60 min of duration, which starts with a 10 min warm-up and are completed with a meditation/relax session.
  Arms: Standard of Care (SOC) + strength training

SUMMARY:
The scope of the STRONG_2 project is to investigate the effect of supervised exercise as add-on to standard of care (SOC), for patients with eating disorders (EDs). The effect of supervised strength training will be measured on health parameters such as muscle strength. The study includes patients diagnosed with anorexia nervosa and in treatment at the Mental Health Center Ballerup (PCB) in the Capital Region of Denmark.

DETAILED DESCRIPTION:
Eating disorders (EDs) are the most common psychiatric disorder affecting young women and contribute with serious psychological, social, physical health complications, and a high mortality rate.

The first general treatment goal of EDs is to address medical complications and suicide risk, and then pathological health effects of the EDs such as bingeing and vomiting. Thereafter, the aim is to address ED psychopathology and behaviors via different forms of psychotherapy. Medical treatment is also used to treat comorbidities.

Treatment of EDs using standard of care (SOC) often implies a reduction in physical activity, and exercise is often prohibited during the intense phase of weight restoration. Since many patients for lengthy periods of time use excessive exercise as a way of compensatory behavior for calorie intake, the sudden stop in physical activity may trigger anxiety and lack of compliance during the weight restoration program. In addition, many ED patients have osteopenia, reduced muscle mass and show signed of depressiveness, all of which benefits from physical activity.

In order to change unhealthy exercise in patients with eating disorders, it may be beneficial to experience exercise in a novel way as part of the treatment for EDs. The number of studies describing supervised exercise for patients with EDs are few, especially for studies examining the effects of implementing exercise in the treatment of EDs in a Danish context. The National Clinical Guidelines suggest that supervised physical activity should be considered in the weight gaining phase as a supplement for common treatment for patients with anorexia nervosa (AN), although there is no description of how this intervention should be implemented (Sundhedsstyrelsen 2005). Knowledge concerning patients' pathological use of training and how this could be managed during rehabilitation is inadequate.

The STRONG_2 project will compare the effects of supervised strength training as add on to standard of care (SOC) vs. SOC alone, in patients with EDs at the Mental Health Center Ballerup (PCB) in the Capital Region of Denmark. Training effects on health parameters including muscle strength, eating disorder psychopathology and pathological exercise will be explored.

The STRONG_2 study will enable an increased understanding of the effects of supervised strength training on muscle strength, increase in muscle mass, and improved bone health, metabolism as well as ED psychopathology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AN according to the International Classification of Disorders version 10 (ICD-10)
2. Age 18-35
3. BMI > 14.5
4. Signed informed consent form-

Exclusion Criteria:

1. Forced care
2. Unstable medical or psychiatric health
3. Issues with compliance to treatment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Maximal strength leg press | Base line, week 6, week 12
  Difference in muscle strength measured with leg press strength tests in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Strength test measurement tool is leg press measured with 1 repetition maximum (1RM) in Kilograms (kg).
Maximal strength bench press | Base line, week 6, week 12
  Difference in muscle strength measured with bench press strength tests in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Strength test measurement tool is bench press measured with 1 repetition maximum (1RM) in Kilograms (kg).
Maximal strength pull down | Base line, week 6, week 12
  Difference in muscle strength measured with pull down strength tests in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Strength test measurement tool is pull down measured with 1 repetition maximum (1RM) in Kilograms (kg).

SECONDARY OUTCOMES:
EDI-DT subscale score | Baseline, week 6, week 12, week 24
  Difference in drive for thinness measured with EDI questionnaire scores in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 1 to 6 where 6 means a better outcome.
EDI subscale score | Baseline, week 6, week 12, week 24
  Difference in body dissatisfaction measured with EDI questionnaire scores in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 1 to 6 where 6 means a better outcome.
Changes in Eating Disorder Symptoms | Baseline, week 12, week 24
  Difference in eating disorder symptoms measured with EDE-Q questionnaire in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 0 to 6 where 6 means a worse outcome.
VAS-mood | Baseline, week 1, week 6, week 12, week 24
  Difference in mood measured with VAS-mood in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a Vas-scale from 0 to 10. For anxiety 10 means a worse outcome, for behavior 10 means a worse outcome and for feelings 10 means a worse outcome and for a happiness question 10 means the best outcome.
Anxiety (HAM-A-6) | Baseline, week 6, week 12, week 24
  Difference in anxiety measured with HAM-A-6 questionnaire in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 0 to 4 and higher total score means a worse outcome.
ERQ total score | Baseline, week 6, week 12, week 24
  Difference in emotional reactivity measured with ERQ questionnaire total score in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 1 to 7. With respect to questions for Cognitive Reappraisal Facets a higher score means better outcome and for questions regarding Expressive Suppression Facets a higher score means a worse outcome.
RMR assessed by indirect calorimetry (ventilated open hood) and RMRratio | Baseline, week 6, week 12
  Difference in resting metabolic rate measured with indirect calorimetry and RMRratio in patients treated with standard of care alone compared to patients treated with standard of care and strength training.
BMD assessed by Dual-energy X-ray Absorptiometry (DXA) | Baseline, week 12
  Difference in bone mineral density measured by Dual-energy X-ray Absorptiometry (DXA) (total bone mineral content, BMD lumbar spine and femur neck[g/m2]) in patients treated with standard of care alone compared to patients treated with standard of care and strength training.
Anthropometry | Baseline, week 12
  Difference in anthropometry (bodyweight, fat mass, and fat free mass) measured with DXA in patients treated with standard of care alone compared to patients treated with standard of care and strength training.
Blood samples Lipid profiles | Baseline,week 12
  Difference in biological parameters measured by changes in lipid levels, like cholesterol, high-density lipoprotein, low-density lipoprotein, very-low-density lipoproteins, triglycerides, free fatty acids, apolipoprotein a1 and B in blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training. Lipidomics, a mass spectrometry based systems level analysis of lipids will be applied for level analysis of lipids and their interacting partners. High or low risk lipid-profiles will be analysed in the two patient groups with high risk lipid profiles expected to mean a worse outcome.
Blood samples Hormones | Baseline,week 12
  Difference in biological parameters measured by changes in hormone levels, like insulin, prostaglandins, cortisol, follicle stimulating hormone, ghrelin, obestatin, resistin, des- acyl-ghrelin, acyl-ghrelin, growth hormone, oxytocin, T3, cortisol, IGF-1, prolactin, estrogen, 17-beta-estradiol, LH, adiponectin, leptin, agouti-related protein, cholecystokinin, alpha-MSH, as well as related variants in blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training.
  The project will examine whether higher levels or lower levels are correlated with a worse or better outcome in the two patient groups.
Blood samples Neuronal biomarkers | Baseline,week 12
  Difference in biological parameters measured by changes in neuronal biomarker levels, like Glial cell line derived neurotrophic factor, Brain derived neurotrophic factor, Wnt- signaling pathway, nerve growth factor, insulin-like growth factor, S-110b, Neuron specific enolase, monoamines as well as related metabolites/variants, neuropeptide Y, HMGB1, as well as related isoforms in blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training.
  The project will examine whether higher levels or lower levels are correlated with a worse or better outcome in the two patient groups.
Weekly binge eating | Baseline, week 1,2,3,4,5,6,7,8,9,10,11,12 and week 24
  Difference in weekly binge eating noted every week of the study in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured as number of binge eating during the week. A higher score means a worse outcome.
Vomiting | Baseline, week 1,2,3,4,5,6,7,8,9,10,11,12 and week 24
  Difference in weekly vomiting noted every week of the study in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured as number of vomiting during the week. A higher score means a worse outcome.
Weekly use of laxatives | Baseline, week 1,2,3,4,5,6,7,8,9,10,11,12 and week 24
  Difference in weekly use of laxatives noted every week of the study in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured as number of laxative use per week and the dose of the specific laxative used. A higher score and dose per week means a worse outcome.
EAI score | Baseline, week 6, week 12, week 24
  Difference in exercise addiction measured with (Exercise Addiction Inventory) EAI score in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured on a scale from 1 to 5 where higher score means a worse outcome.
EDS score | Baseline, week 6, week 12, week 24
  Difference in exercise addiction measured with Exercise Dependence Scale (EDS) score in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured on a scale from 1 to 6 where higher score means a worse outcome.
Body Awareness test (BAT) | Baseline, week 1,2,6,7,12 and week 24
  Difference in body awareness measured with Body Awareness test (BAT) in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Questions are scored on a scale ranging from never to always with four items in between. Always means a worse outcome except for two questions regarding body satisfaction and relaxation where always means a better outcome.
Compulsive Exercise test | Baseline, week 1, 2, 6, 7, 12 and week 24
  Difference in compulsive exercise measured with Compulsive Exercise test (CET) in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured on a scale from 0 to 5 where higher score means a worse outcome except for two questions where higher score means better outcome.
Activity and sleep tracking via Actigraph | Baseline, week 6, week 12, week 24
  Difference in activity/sleep measured with Actigraph in patients treated with standard of care alone compared to patients treated with standard of care and strength training.
Readiness and motivations interview | Baseline, week 1, week 6, week 7, week 12, week 24
  Difference in readiness/motivations measured with Readiness and motivations interview in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured on a scale from 1 to 10 where higher score means a better outcome.
Patient satisfaction: Expectations and experiences of ED-treatment scale | Baseline, week 6, week 12, week 24
  Difference in patient satisfaction measured with the Expectations and experiences of ED-treatment scale (Clinton 2001) in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 0 to 2 where higher score means worse outcome.
Global Assessment of Functioning (GAF) | Baseline, week 6, week 12, week 24
  Difference in social functioning measured with numeric scale using the Global Assessment of Functioning (GAF-F and GAF-S) in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is measured on a scale from 1 to 99 where lower score means a worse outcome.
Clinical Global Impression (CGI) | Baseline, week 6, week 12, week 24
  Difference in severity of the patient's illness measured with 7-point scale using the Clinical Global Impression - Severity scale (CGI-S) in patients treated with standard of care alone compared to patients treated with standard of care and strength training. Scoring is on a scale from 1 to 7 where higher score means worse outcome.
Bone turnover CTX-1 | Baseline, week 12
  Difference in bone turnover measured with analyses of the bone marker CTX-1 from blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training. High levels above reference range which is 50 - 450 measured in pg/ml indicate worse outcome.
Bone turnover PN1P | Baseline, week 12
  Difference in bone turnover measured with analyses of the bone formation marker PN1P from blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training. High levels above normal reference range which is 20 - 85 measured in microgram/L can indicate worse outcome.
Bone turnover Osteocalcin | Baseline, week 12
  Difference in bone turnover measured with analyses of the bone marker Osteocalcin from blood material from patients treated with standard of care alone compared to patients treated with standard of care and strength training. Increased levels above normal reference range which is 0.7 - 6.5 measured in ng/ml mean higher osteoblast activity and formation of new bone and mean better outcome for most patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Magnus Sjögren, MD, PhD, Principal Investigator — Eating disorder unit, Mental Health Services in the Capital Region, Ballerup; Louise B Rasmussen, MD, PhD, Study Chair — Mental Health Services in the Capital Region, Ballerup
Locations (2):
- Denmark (2):
  - Eating disorder unit, Mental Health Center, Ballerup Municipality, Danmark
  - Institut for Idræt og Ernæring, NEXS, University of Copenhagen, Copenhagen